CLINICAL TRIAL: NCT00899210
Title: Study of Diagnostic Tests Studying Kinetic Variation of Serum Matrix Metalloproteases After Surgical Treatment and/or Destruction by Radiofrequency in Patients With Hepatic Metastases From Colorectal Cancer
Brief Title: Matrix Metalloproteinases After Surgery and/or Radiofrequency Ablation in Patients With Liver Metastases From Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000574192; CHUG-METALLO-1; RECF0455
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; adenocarcinoma of the colon; stage IV colon cancer; adenocarcinoma of the rectum; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Cryosurgery; Radiofrequency Ablation

INTERVENTIONS:
Other: laboratory biomarker analysis
Procedure: cryosurgery
Procedure: radiofrequency ablation
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research trial is studying matrix metalloproteinases after surgery or radiofrequency ablation in patients with liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Describe the kinetics of postoperative changes of serum matrix metalloproteinases (MMP) (MMP-1, MMP-2, MMP-7, MMP-9) and their inhibitors (TIMP) (TIMP-1, TIMP-2) as a function of surgical technique.

Secondary

* Determine the predictive value of postoperative risk of recurrence.
* Correlate the risk of recurrence with surgical technique.
* Determine whether elevated serum levels of MMP are a better marker than the carcinoembryonic antigen of hepatic or extrahepatic recurrence.
* Determine whether the postoperative serum of HGF/SF is correlated to changes in plasma levels of MMPs.

OUTLINE: Blood samples are collected periodically before and after treatment to analyze for metalloproteinases and their inhibitors.

After completion of study treatment, patients are followed at day 45 and then every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Patients with histologically confirmed adenocarcinoma of the colon or rectum and liver metastases

    * Must have undergone prior complete resection of the tumor more than 3 months ago
    * Liver metastases must be resectable or accessible for radiofrequency ablation
  * Patients undergoing cryosurgery of the digestive tract for a reason other than cancer or infection (control)

PATIENT CHARACTERISTICS:

* No other neoplastic disease that is measurable or being treated other than colorectal cancer
* No heart failure or severe respiratory disease
* No uncontrolled infection or other severe disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No participation in another study involving new drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2003-09; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Kinetics of postoperative changes of serum matrix metalloproteinases (MMP) and their inhibitors (TIMP)

SECONDARY OUTCOMES:
Predictive value of postoperative risk of recurrence
Correlation of risk of recurrence with surgical technique
Elevated serum levels of MMP vs carcinoembryonic antigen as a marker of hepatic or extrahepatic recurrence
Correlation of postoperative serum HGF/SF with plasma levels in MMPs

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rebischung, Study Chair — University Hospital, Grenoble